CLINICAL TRIAL: NCT05455957
Title: The Effect of Neuromuscular and Vestibulo-Ocular Reflex Training Program on Balance, Isokinetic Muscle Strength and Proprioception in Subjects With Chronic Ankle Instability
Brief Title: The Effect of Neuromuscular and Vestibulo-Ocular Training on Balance,Isokinetic Strength and Proprioception in Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YeditepeU1
Record Dates: First submitted 2022-06-10; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Chronic Ankle Instability
Keywords: ankle instability, balance, neuromuscular,vestibulo-ocular
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training (Experimental): The neuromuscular exercise training group includes single-leg stance, single leg hop and strength exercise.Each training session took approximately 60 minutes and 3 times a week for 4 weeks.The neuromuscular group included supervised, strength, balance and hop stabilization exercises on the different surfaces that focus on the restoring of static and dynamic balance. Both groups completed strength exercises in the same way. Strength exercises include ;4-way ankle theraband exercises,foot intrinsic strengthening (toe curl, doming),heel raises exercise,squat, lunge activities.Balance exercises include single-leg stance single leg hop and unticipated hop to stabilization activities.
  Interventions: Other: exercise
- Vestibulo-Ocular Reflex Training (Experimental): The vestibulo ocular reflex training group includes head and gaze stability exercises in addition to single le stance,single leg hop and strength exercise.Each training session took approximately 60 minutes and 3 times a week for 4 weeks.In the vestibulo- ocular exercise program, individuals tried to maintain their balance with head and eye movements in addition to balance and hop stabilization activities. Both groups completed strength exercises in the same way. Strength exercises include ;4-way ankle theraband exercises,foot intrinsic strengthening (toe curl, doming),heel raises exercise,squat, lunge activities.Balance exercises include single-leg stance single leg hop and unticipated hop to stabilization activities.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — neuromuscular and vestibulo-ocular training

SUMMARY:
The aim of the study is to compare the effects of neromuscular exercise combined with vestibulo-ocular reflex training on balance,isokinetic muscle strength and proprioception in subjects with ankle instability.The aim of the study is to compare the effects of neromuscular exercise combined with vestibulo-ocular reflex training on balance and isokinetic muscle strength in subjects with ankle instability.

Hypotheses of the study; H0: Vestibulo-ocular reflex training protocol, which is given in addition to the neuromuscular exercise program, has an effect on isokinetic ankle muscle strength and balance in individuals with ankle instability.

H1: Vestibulo-ocular reflex training protocol, which is given in addition to the neuromuscular exercise program, has no effect on isokinetic ankle muscle strength and balance in individuals with ankle instability.

DETAILED DESCRIPTION:
The aim of the study is to compare the effects of neromuscular exercise combined with vestibulo-ocular reflex training on balance,isokinetic muscle strength and proprioception in subjects with ankle instability. This study was conducted in Sportomed Athlete Health and Orthopedic Rehabilitation clinic in February 2020, September 2022.A total of 20 participants aged 18-30 were included in the study on a voluntary basis..Participants were randomly seperated to 2 groups. Demographic information and informed consent forms were filled into all subjects who volunteered to participate in the study and in accordance with the research criteria. After the evaluation, the subjects in the first group were included in the vestibulo-ocular exercise program in addition to the neuromuscular exercise programs with the same physiotherapist. Subjects in the second group were included in neuromuscular training programs. The trainings were applied three days a week for four weeks and each training session lasted approximately 60 minutes. Functional limitations of the participants before and after the treatment were evaluated with the Foot and Ankle Ability Measure Daily Living Subscale (FAAM-ADL) and Sports Subscale (FAAM-S). Dynamic balance evaluation with star excursion balance test, proprioception evaluation by measuring joint position sense with goniometer, and ankle evertor and inverter concentric muscle strength were evaluated using isokinetic dynamometer at angular velocities of 60/s, 120/s and 180/s, and the results were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-30 years old
* At least 2 lateral sprains to the same ankle in the past
* At least 1 episode of "giving way" that had occurred within the past 6 months
* The presence of residual symptoms during functional activities and had to be free from symptoms of any other previous injury to the lower extremity.
* No other injuries to the lower limbs

Exclusion Criteria:

* Having a bilateral ankle instability
* Having a history of ankle fracture
* Having a history of fracture or surgery to the involved lower extremity
* Having a history of balance and vestibular disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
balance,isokinetic muscle strength,proprioception | 1 hours
  Dynamic balance evaluation with star excursion balance test recorded in centimeters.
isokinetic muscle strength | 1 hours
  ankle evertor- inverter concentric muscle strength by using isokinetic dynamometer at angular velocities of 60 degree/s, 120 degree /s and 180 degree/s were recorded.
proprioception | 1 hours
  Proprioception was evaluated by measuring joint position sense with a goniometer, and deviations in proprioception were recorded as degrees.

SECONDARY OUTCOMES:
weight | 1 hours
  kilogram
height | 1 hours
  meter

CONTACTS AND LOCATIONS:
Locations (1):
- Sportomed, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided